CLINICAL TRIAL: NCT06226831
Title: Onset of Lower Urinary Tract Symptoms in Multiple Sclerosis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: MS001
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Lower Urinary Tract Symptoms; Multiple Sclerosis
Keywords: Multiple Sclerosis; Lower-Urinary Tract Symptoms; Urinary Urgency; Cerebellar and/or Pyramidal Symptoms
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS with LUTS: Patients with multiple sclerosis with LUTS symptoms.
  Interventions: Other: Structured interview
- MS without LUTS: Patients with multiple sclerosis without LUTS symptoms.
  Interventions: Other: Structured interview

INTERVENTIONS:
Other: Structured interview — In-person structured interviews will be performed by the investigators.

SUMMARY:
Retrospective, non-interventional case-control study, the patients were asked about their first lower-urinary tract symptoms and the date of their onset, using a structured interview. The information was matched with the medical records.

DETAILED DESCRIPTION:
This retrospective non-interventional case-control study will be conducted at a single tertiary referral Multidisciplinary Centre for Diagnostics and Treatment of MS at the University Hospital, Ostrava, Czech Republic. The study will be performed per the Declaration of Helsinki, World Health Organization. The study protocol has been approved by the Ethics Committee of University Hospital Ostrava, Nr.289/19.

The database of the Center includes medical records of all consecutive patients, who have visited the center at least once, starting from 1996 until the present day. Based on the inclusion criteria of proven multiple sclerosis (MS) diagnosis and the current age over 18 years, the initial database search identified eligible 2348 individuals. During the routine follow-up visit of the patients at the Center, a structured in-person interview led by a physician will be performed.

The data from this interview will be cross-checked with the medical records. In addition to standard demographic variables, the following data will be obtained:

Age 1 - Age at the onset of the first symptoms of MS Age 2 - Age at the time of diagnosis of MS Age 3 - Age at the time of data collection MS course - patients with a primary progressive, secondary progressive, or progressive relapsing disease at the time of data collection will be included in the group "Progressive MS course". The "Relapsing-remitting MS course" group will include patients who had a relapsing-remitting disease and those with isolated clinical symptoms at the time of data collection.

CPS - The "CPS yes" group will include patients who experienced cerebellar and/or pyramidal symptoms (CPS) as the first manifestation of MS. Patients with other first manifestations, such as optic neuritis, sensory disturbances, etc., will be included in the "CPS no" group.

OCB - The "OCB yes" group will include patients with oligoclonal bands (OCB) in the cerebrospinal fluid at the time of diagnosis of MS. Patients in whom OCB in the cerebrospinal fluid at the time of diagnosis of MS will not be identified, will be assigned to the "OCB no" group.

LUTS - The "LUTS yes" group will include patients with the presence of at least one LUTS at the time of the structured interview. In this group, a complete list of LUTS with layman descriptions will be given to each patient. The patients will be asked to indicate, which of the lower urinary tract symptoms (LUTS) occurred as the very first one. The "LUTS no" group will include patients without LUTS.

EDSS 1 - The Expanded Disability Status Scale (EDSS) total score will be collected after stabilization following the first MS relapse before the disease-specific treatment will be initiated, and will be defined as the baseline EDSS at the time of MS diagnosis.

EDSS 2 - EDSS at the time of first onset of LUTS. D1- duration of MS symptoms, i.e. time elapsed since the onset of first symptoms attributable to MS.

D2 - MS disease duration, i.e. the time elapsed since the diagnosis of MS will be determined.

D3 - duration of LUTS, i.e. the time elapsed since the first LUTS appeared.

Based on the above-mentioned data, collected during the interview, the researchers will calculate the following variables:

T1 - Time between the presentation of first symptoms attributable to MS and the onset of first LUTS (T1= D1-D3) T2 -Time between the diagnosis of MS and the onset of first LUTS (T2= D2-D3)

Based on LUTS presence and its relationship to the time of diagnosis of MS, the patients will be divided into 3 groups:

Group A - Patients in whom LUTS appeared after the first neurological symptom which could be attributed to the MS has developed and diagnosis of MS was established; Group B - Patients who have not developed LUTS yet; Group C - Patients in whom LUTS appeared before the diagnosis of MS was established.

STATISTICAL ANALYSIS Numerical variables will be expressed as the median and the interquartile range. Categorical variables will be presented as the absolute frequencies and relative frequencies in percentages. Defined groups will be compared using the Mann-Whitney test, the Kruskal-Wallis test, or the Chi-square test of independence for contingency tables. The first two mentioned tests will be also used to test the difference between other subgroups of interest. The statistical dependence of two numerical variables will be tested and evaluated using Spearman's rank correlation coefficient and its test of significance. The univariate logistic regression will be used to assess the significance of selected factors in relation to the development of LUTS. The results will be presented with the odds ratios and corresponding confidence intervals and will be visualized using the forest plot. Finally, the methods of survival analysis - the Kaplan-Meier curve and the Cox proportional-hazards model, will be used for the analysis of survival without LUTS. All statistical analyses will be performed using R software (version 4.0.2, www.r-project.org) and the significance level will be set to 0.05.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of multiple sclerosis
* adult patients
* signed informed consent

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with the diagnosis of MS, with or without LUTS.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
LUTS onset | 1 hour of structured interview
  The time of LUTS onset in relation to the diagnosis of MS diagnosis (before or after) will be observed in months, during the structured interviews with the study subjects.

SECONDARY OUTCOMES:
Course of disease (clinical examination) | 5 years
  The course of disease (primary-progressive, secondary-progressive) will be observed, defined by the presence or absence of cerebro-pyramidal symptoms (YES/NO - defined with clinical examination).
Course of disease (EDSS scale) | 5 years
  The course of disease (primary-progressive, secondary-progressive) will be observed, defined by the presence or absence of cerebro-pyramidal symptoms (defined by the Kurtzke Expanded Disability Status Scale (EDSS)). The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Krhut, prof.,MD, PhD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make the individual participant data available to other researchers. The data may be provided upon request.

REFERENCES:
- [Background] Dilokthornsakul P, Valuck RJ, Nair KV, Corboy JR, Allen RR, Campbell JD. Multiple sclerosis prevalence in the United States commercially insured population. Neurology. 2016 Mar 15;86(11):1014-21. doi: 10.1212/WNL.0000000000002469. Epub 2016 Feb 17. PMID 26888980
- [Background] Rosati G. The prevalence of multiple sclerosis in the world: an update. Neurol Sci. 2001 Apr;22(2):117-39. doi: 10.1007/s100720170011. PMID 11603614
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Nortvedt MW, Riise T, Myhr KM, Landtblom AM, Bakke A, Nyland HI. Reduced quality of life among multiple sclerosis patients with sexual disturbance and bladder dysfunction. Mult Scler. 2001 Aug;7(4):231-5. doi: 10.1177/135245850100700404. PMID 11548982
- [Background] Khalaf KM, Coyne KS, Globe DR, Malone DC, Armstrong EP, Patel V, Burks J. The impact of lower urinary tract symptoms on health-related quality of life among patients with multiple sclerosis. Neurourol Urodyn. 2016 Jan;35(1):48-54. doi: 10.1002/nau.22670. Epub 2014 Oct 18. PMID 25327401
- [Background] Khalaf KM, Coyne KS, Globe DR, Armstrong EP, Malone DC, Burks J. Lower urinary tract symptom prevalence and management among patients with multiple sclerosis. Int J MS Care. 2015 Jan-Feb;17(1):14-25. doi: 10.7224/1537-2073.2013-040. PMID 25741223
- [Background] Al Dandan HB, Coote S, McClurg D. Prevalence of Lower Urinary Tract Symptoms in People with Multiple Sclerosis: A Systematic Review and Meta-analysis. Int J MS Care. 2020 Mar-Apr;22(2):91-99. doi: 10.7224/1537-2073.2019-030. PMID 32410904
- [Background] Lublin FD, Reingold SC, Cohen JA, Cutter GR, Sorensen PS, Thompson AJ, Wolinsky JS, Balcer LJ, Banwell B, Barkhof F, Bebo B Jr, Calabresi PA, Clanet M, Comi G, Fox RJ, Freedman MS, Goodman AD, Inglese M, Kappos L, Kieseier BC, Lincoln JA, Lubetzki C, Miller AE, Montalban X, O'Connor PW, Petkau J, Pozzilli C, Rudick RA, Sormani MP, Stuve O, Waubant E, Polman CH. Defining the clinical course of multiple sclerosis: the 2013 revisions. Neurology. 2014 Jul 15;83(3):278-86. doi: 10.1212/WNL.0000000000000560. Epub 2014 May 28. PMID 24871874
- [Background] KURTZKE JF. A new scale for evaluating disability in multiple sclerosis. Neurology. 1955 Aug;5(8):580-3. doi: 10.1212/wnl.5.8.580. No abstract available. PMID 13244774
- [Background] Medina-Polo J, Adot JM, Allue M, Arlandis S, Blasco P, Casanova B, Matias-Guiu J, Madurga B, Meza-Murillo ER, Muller-Arteaga C, Rodriguez-Acevedo B, Vara J, Zubiaur MC, Lopez-Fando L. Consensus document on the multidisciplinary management of neurogenic lower urinary tract dysfunction in patients with multiple sclerosis. Neurourol Urodyn. 2020 Feb;39(2):762-770. doi: 10.1002/nau.24276. Epub 2020 Jan 15. PMID 31943361
- [Background] Krhut J, Hradilek P, Zapletalova O. Analysis of the upper urinary tract function in multiple sclerosis patients. Acta Neurol Scand. 2008 Aug;118(2):115-9. doi: 10.1111/j.1600-0404.2008.00992.x. Epub 2008 Feb 25. PMID 18307573
- [Background] Phe V, Pakzad M, Curtis C, Porter B, Haslam C, Chataway J, Panicker JN. Urinary tract infections in multiple sclerosis. Mult Scler. 2016 Jun;22(7):855-61. doi: 10.1177/1352458516633903. Epub 2016 Feb 18. PMID 26892318
- [Background] Correale J, Fiol M, Gilmore W. The risk of relapses in multiple sclerosis during systemic infections. Neurology. 2006 Aug 22;67(4):652-9. doi: 10.1212/01.wnl.0000233834.09743.3b. Epub 2006 Jul 26. PMID 16870812